CLINICAL TRIAL: NCT01999439
Title: Quantitative MRI Evaluation of Esophageal Remodeling/Response to Treatment in Children and Adolescents With Eosinophilic Esophagitis Presenting With Dysphagia
Brief Title: EoE(Eosinophilic Esophagitis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ethan Smith, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00080065
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Eosinophilic Esophagitis; Dysphagia
MeSH Terms: conditions — Eosinophilic Esophagitis; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eosinophilic Esophagitis with Dysphagia (Experimental): To assess quantitative magnetic resonance imaging(MRI)as a potential diagnostic tool for evaluating esophageal wall thickness and stiffness and response to treatment in children and adolescents with a diagnosis of eosinophilic esophagitis (EoE) presenting with difficulty swallowing(dysphagia)and food impaction.
  Interventions: Procedure: Eosinophilic Esophagitis with Dysphagia

INTERVENTIONS:
Procedure: Eosinophilic Esophagitis with Dysphagia — An upper endoscopy with biopsy at the time of diagnosis(which is a standard procedure to diagnose eosinophilic esophagitis. This will be done with sedation or general anesthesia, also a standard procedure. At the time of the anesthesia a small amount of blood will be drawn to measure markers of inflammation and fibrosis. This procedure will take approximately 45 minutes to complete. This endoscopy with biopsy will be repeated in 6 months.
  Subjects will also complete a magnetic resonance imaging(MRI)scan with 2 weeks of the initial clinical endoscopy with biopsy, prior to the initiation of your medical treatment. This MRI will be repeated in 6 months. Each magnetic resonance imaging(MRI)scan will take approximately 2 hours to complete.
Procedure: Eosinophilic Esophagitis with Dysphagia — Subjects will also complete a magnetic resonance imaging(MRI)scan with 2 weeks of the initial clinical endoscopy with biopsy, prior to the initiation of your medical treatment. This MRI will be repeated in 6 months. Each magnetic resonance imaging(MRI)scan will take approximately 2 hours to complete.

SUMMARY:
To evaluate quantitative magnetic resonance imaging(MRI) as a potential non-invasive, radiation-free diagnostic tool for evaluating esophageal wall remodeling (thickness and stiffness) and response to treatment in children and adolescents with newly diagnosed eosinophilic esophagitis (EoE) presenting with dysphagia (difficulty swallowing) and food impaction.

DETAILED DESCRIPTION:
Eosinophilic esophagitis(EoE) is a form of chronic inflammation affecting the esophagus which often results in wall thickening and esophageal stiffening and is associated with complications, such as esophageal tears and strictures (narrowings). Chronic dysphagia and acute food impaction (swallowed food stuck in the esophagus) are common symptoms of EoE and are associated with esophageal wall thickening and stiffness.

Current diagnostic techniques such as endoscopy with biopsy give only limited information about changes in the esophageal wall in eosinophilic esophagitis(EoE). In routine clinical practice, repeat endoscopic evaluation with biopsy is commonly performed about 3-6 months after initial therapy for eosinophilic esophagitis(EoE). However, follow-up endoscopy with biopsy has drawbacks as it is invasive, costly and typically requires deep sedation or general anesthesia.

We propose to evaluate quantitative MRI as a potential non-invasive diagnostic option for evaluating esophageal wall remodeling in patients with eosinophilic esophagitis(EoE).

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients ages 8 to 18 years of age.
2. Pediatric patients with dysphagia(difficulty swallowing) or an episode of food impaction.
3. Pediatric patients newly diagnosed with Eosinophilic Esophagitis -

Exclusion Criteria:

1. Are not able to undergo an MRI without needing sedation or general anesthesia
2. Are allergic to gadolinium-based contrast material
3. Have an ongoing acute kidney injury
4. Have chronic kidney disease with an estimated glomerular filtration rate(eGFR)of <40 ml/min.
5. Have a presence of eosinophilia involving the stomach and/or esophagus.
6. Have a prior history of caustic ingestion
7. Have a prior history of esophageal surgery, including history of tracheoesophageal fistula.
8. Have known celiac disease
9. Have known Crohn's disease
10. Have known malignancy
11. Have hypereosinophilic syndrome
12. Have recent history of parasitic infection
13. Have known inflammatory bowel disease -

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of quantitative MRI as a diagnostic option for eosinophilic esophagitis | 2 years
  To assess noninvasive quantitative magnetic resonance imaging (MRI) based biomarkers in the evaluation of esophageal wall remodeling and response to treatment in children and adolescents with newly diagnosed eosinophilic esophagitis presenting with dysphagia. Magnetic resonance imaging (MRI)findings will be correlated with the endoscopic appearance of the esophagus, histologic findings, and clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Smith, M.D., Principal Investigator — C.S. Mott Childrens Hospital
Locations (1):
- University of Michigan C. S. Mott Childrens Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No